CLINICAL TRIAL: NCT05125484
Title: Comparison Of Bowen's Technique And Myofascial Release Technique On Pain And Disability In Patients With Trapezitis
Brief Title: Comparison of Bowen's Technique and Myofascial Release Technique On Pain And Disability in Trapezitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RiphahIU Zainab Rana
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Trapezius Muscle Strain
Keywords: Bowen therapy; Myofacial Release Technique; Isometric Scapular pinch test; Lateral Scapular Slide test; NDI

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Intervention group 1 (Experimental): Patient was in lying position. Therapist placed thumb on the effected side muscke. Then hooked thumb on lateral edge of muscle to apply pressure against the muscle. Took a pause. Thumb flattened in a medial direction and pluck was created in muscle.
  Set of 15-20 bowen moves on upper , middle and lower fibres each with 2 mins gap between each set.
  Total treatment time: 20 mins
  Interventions: Other: experimental Bowen Technique
- Experimental interventional group II (Experimental): Patient was in lying position. MFR applied via ulnar border of both palms while patient being in contralateral side flexion.
  20 mins
  Interventions: Other: Experimental Myofacial release technique

INTERVENTIONS:
Other: experimental Bowen Technique — Patient was in lying position. Therapist placed thumb on the effected side muscke. Then hooked thumb on lateral edge of muscle to apply pressure against the muscle. Took a pause. Thumb flattened in a medial direction and pluck was created in muscle.
  Set of 15-20 bowen moves on upper , middle and lower fibres each with 2 mins gap between each set.
  Total treatment time: 20 mins
  Arms: Experimental Intervention group 1
Other: Experimental Myofacial release technique — Patient was in lying position. MFR applied via ulnar border of both palms while patient being in contralateral side flexion.
  20 mins
  Arms: Experimental interventional group II

SUMMARY:
The aim of this research is to compare the effects of Bowen's technique and Myofascial Release technique on pain and disability in patients with trapezitis.Randomized controlled trials done at Islamabad Physiotherapy and Rehabilitation Centre(IPRC) and Benazir Bhutto Hospital. The sample size was 66. The subjects were divided in two groups, 33 subjects in Bowen's Technique group and 33 subjects in Myofascial Release Technique group. Study duration was of 6 months. Sampling technique applied was non probability purposive sampling technique. The patients aged 20-40 years and clinicaly diagnosed with Trapezitis(spasm,trigger points,tenderness,stiffness) were included in the study. Tools used in the study are Cervical ROMs, NPRS, NDI, Isometric Scapular Pinch Test and Lateral Scapular Slide Test.

DETAILED DESCRIPTION:
Trapezitis is a condition that involves inflammation of the trapezius muscle. The upper fibers of trapezius, being the postural muscles, are highly susceptible to overuse injuries and thus the inflammation.This results in pain that is present during the rest, is aggravated with activity and is referred to the other areas. The pain results in protective spasm of the antagonistic muscle group that also restricts the passive range of motion and makes it painful too. In people working for long hours at a desk and computers or spending many hours driving, the low level of upper trapezius activity is frequently found because of head posture during sitting and standing , which is common cause of tension and neck pain in such people.Various recent studies have hypothesized that trapezitis occurs due to muscle tissue overloading and injury, that results in involuntary shortening of localized muscle fibers. The stressed soft tissue area thus receives less glucose, oxygen and nutrients supply; subsequently high levels of metabolic waste products are accumulated. And this cascade of events ends in altered status of tissue, pain and the development of the Trigger points in the muscle.

Myofascial Release(MFR) is a soft tissue mobilization technique that is defined as " the facilitation of mechanical, neural and psycho physiological adaptive potential as interfaced via the myofascial system".MFR decreases the pain and restores the proper alignment by changing the ground substance's viscosity to more fluid state resulting in elimination of excessive pressure of fascia on the pain sensitive structures.

There is one more soft tissue technique called 'Bowen Technique' that is useful and indicated in myofascial pain. The Bowen technique is defined as:

'…dynamic system of muscle and connective tissue therapy which balances the body to allow it to heal itself. The work consists of a series of precise moves on specific points of the body. These moves are light and can be done through clothing. There are frequent and important pauses between each series of moves giving the body time to benefit from each. The technique uses positive moves that initiate a positive energy flow and negative moves that isolate this energy to a specific area' (Rentsch and Rentsch,1997) The Bowen technique was developed by late Tom Bowen in Geelong, Australia in 1950. It is a connective tissue technique that uses subtle inputs called 'Bowen moves' to the body that stimulates the body's self-healing. The Bowen moves applied are in several sets in a complete session of 15-45 minutes duration. While applying the technique, the therapist uses the thumb when the Bowen move is executed away from the patient's body and two fingers are used when the Bowen move is executed towards the patient's body. The technique can be used anywhere on the origin, insertion or the belly of the muscle and produces a physical and an energetic action.

This technique can be used to treat many types acute and chronic injuries and other health issues. It does this by using holistic approach in which body's innate healing mechanism is stimulated. This technique has been recommended in many conditions like headache, cervical pain, back pain, whiplash injury, TMJ dysfunction, herniated disk, tennis elbow, hamstring tightness and frozen shoulder, work related injuries etc.

An RCT was done by Ekta S. Chaudhary, Nehal Shah, Neeta Vyas, Ratan Khuman1, Dhara Chavda1, Gopal Nambi that compared the effectiveness of MFR and cold pack in Upper trapezius Spasm and concluded both MFR and cold pack along with exercises to be effective in upper trapezium muscle spasm but the overall effects of MFR surpassed the cold therapy. Another study by Pooja Mane , Amrutkuvar Pawar , Trupti Warude compared the effects of Myofascial Release technique with Deep Friction Massage on pain and cervical ROM, the results concluded both therapies to bring improvement in pain and cervical ROM but MFR was more effective. Similarly, a systematic review of RCTs was conducted to determine the effectiveness of MFR in decreasing pain , improving function and elongate length and concluded MFR to be emerging strategy with strong evidence base and solid treatment option for many conditions. A study was conducted to compare the effects of MFR with hot pack in reducing pain and improving passive ROM in shoulder joint and that concluded both to be effective but MFR proved to be more favorable because of the less time spent and no need of equipment.

A study has been done to see the effects of Bowen technique as an adjunct therapy to conventional physiotherapy treatment on the pain and functional outcomes in patient with Acute trapezitis and the results established Bowen technique to be effective in decreasing pain and improving functional outcomes in Acute trapezitis.A few studies were conducted that evaluated the effectiveness of Bowen technique in frozen shoulder and concluded this technique as a positive intervention in improving mobility, functional status and decreasing pain. A few studies were conducted that compared the effects of Bowen technique vs MET in treatment of hamstring tightness.And few other worked to establish the effectiveness of Bowen technique in different complex and common conditions and found positive results.A study was done to show Bowen technique to be effective in health service workplace to improve physical as well as mental well-being of the working staff.

This study aims to compare the short term effects of Bowen Technique and MFR on pain and neck disability in patients with trapezitis. Also it intends to study the short term effects of both techniques on scapular motions. Bowen technique is a relatively new technique, having easier application and has been less worked on. So, if this study proves the effectiveness of Bowen technique in comparison with MFR in patient with trapezitis. Further studies can be conducted to evaluate its efficacy as an independent and preferable procedure in treatment of other conditions and further work can be conducted on other areas as well. As this is a holistic technique, so it could be a beneficial addition in the daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female.
* Age 20-40 years.
* Clinically diagnosed with Trapezitis.(Spasm,stiffness,Tenderness,Trigger Points,Taut band)
* Cummulative trauma disorder
* Occupational overuse syndrome

Exclusion Criteria:

* Any medical conditions or diseases that could interfere with intervention performance.
* Any traumatic neck injury
* Cervical vertebral fracture
* Cervical spinal cord compromise/ cervical myelopathy
* Cervical radiculopathy
* Cervical Spondylolisthesis
* Any tumour
* Any degenerative diseases

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | 3rd day
  It is a 10-item questionnaire each them of having 6 possible answers. The score of each item lies between 0 to 5, where 0 means no pain/ limitation in activities) and 5 means 'as much pain as possible or maximal limitation in activities'.[19] Thus the Total scores range between 0 - 50 points.
Isometric Scapular Pinch Test | 3rd day
  In ISPT the patient actively performs maximal scapular retraction and holds it for 2 seconds. If the pain is present after 15-20 seconds or patient fails to hold it then the test is positive.

SECONDARY OUTCOMES:
Lateral Scapular Slide Test | 3rd day
  LSST is a test that assesses the excessive scapular movement with respect to thoracic spine. A total of three measurements are taken in three positions:
  From scapular spine to T2/T3 level From Inferior scapular angle to T7/T9 level From superior scapular angle to T2 level. Measurments are taken 3 times in 3 positions
NPRS | 3rd day
  pain is measured with the help of numeric pain rating scale that is 11 point scale from 0-10 with 0 referring no pain and 10 represent max pain.
Cervical flexion range of motion | 3rd day
  The range of motion will be measure by goniometer at baseline, after first day treatment and after 3rd day.
Cervical extension range of motion | 3rd day
  The range of motion will be measure by goniometer at baseline, after first day treatment and after 3rd day.
Cervical Rt side flexion range of motion | 3rd day
  The range of motion will be measure by goniometer at baseline, after first day treatment and after 3rd day.
Cervical Lt side flexion range of motion | 3rd day
  The range of motion will be measure by goniometer at baseline, after first day treatment and after 3rd day.
Cervical Rt side Rotation range of motion | 3rd day
  The range of motion will be measure by goniometer at baseline, after first day treatment and after 3rd day.
Cervical Lt side Rotation range of motion | 3rd day
  The range of motion will be measure by goniometer at baseline, after first day treatment and after 3rd day.

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, MSPT-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Benazir Bhutto Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No